CLINICAL TRIAL: NCT01003236
Title: Evaluating the Preventive Effect of Milk Thistle Extract (Silymarin) on Progression of Diabetic Nephropathy, a Randomized, Double-blind, Placebo-controlled Clinical Trial.
Brief Title: Evaluating the Renoprotective Effect of Milk Thistle Extract on Patients With Type II Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ghazal Vessal, Dr, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4774
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; Type II Diabetes; Milk Thistle extract; Silymarin
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — milk-thistle extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): 1 tablet 3 times daily
  Interventions: Drug: placebo
- Milk Thistle extract (Experimental): 1 tablet of the extract (equivalent to 140 mg silymarin) 3 times per day
  Interventions: Drug: Milk Thistle extract

INTERVENTIONS:
Drug: placebo — 140 mg placebo tablets, 3 times per day for 3 months
  Arms: placebo
Drug: Milk Thistle extract — 1 tablet equal to 140mg silymarin administered 3 times a day for 3 months
  Other Names: Livergol made by Goldaru Pharmaceutical Company (Iran)
  Arms: Milk Thistle extract

SUMMARY:
There is considerable evidence that increased blood glucose results in the generation of reactive oxygen species, ultimately leading to increased oxidative stress in a variety of tissues. This may lead to the activation of stress-sensitive intracellular signaling pathways, causing cellular damage and late complications of diabetes including renal injury. Although the investigators understanding of how hyperglycemia-induced oxidative stress ultimately leads to tissue damage has advanced considerably in recent years, effective therapeutic strategies to prevent or delay the development of this damage remain limited. The flavonoid complex silymarin, an extract from the milk thistle, and its major pharmacological active component silibinin are free radical scavengers and potent membrane stabilizers by preventing lipid peroxidation. Furthermore, during early stages of diabetes, flavonoids minimize oxidative stress, and inflammation which represent important factors in the development of diabetic nephropathy.

In this study the investigators plan to evaluate the renoprotective effect of milk thistle extract on type II diabetic patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes
* Overt proteinuria defined by urinary albumin excretion > 300 mg/24 hr in 2 consecutive determinations despite treatment with highest FDA recommended doses of an angiotensin converting enzyme inhibitor or angiotensin receptor blocker for at least 6 months.
* Treatment of hyperglycemia with (but not limited to) an oral hypoglycemic agent or insulin (If a thiazolidinedione is used, stable dose for at least 6 months)
* Treatment of hypercholesterolemia with (but not limited to) one medication from the class statins
* Presence of diabetic retinopathy
* Signing informed consent

Exclusion Criteria:

* Type I diabetes
* Advanced chronic kidney disease defined by estimated GFR < 30 ml/min/1.73 m2
* Severely uncontrolled diabetes defined by HbA1C > 10%
* Uncontrolled hypertension defined by SBP >160 mmHg or DBP >100 mmHg despite antihypertensive therapy
* Secondary forms of hypertension with defined etiology other than diabetes mellitus
* Other renal diseases
* History of solid organ transplantation
* Chronic Heart Failure with NYHA class III or IV
* Active infection
* Pregnancy
* Use of one of the following medications within 2 months prior to enrollment in the study:

  * Non-steroidal anti-inflammatory agents
  * Antioxidants supplements including: vitamin E, vitamin C, N-acetyl- cysteine (NAC), Pentoxyfilline, Lipoic acid, Fish-oil extracts (omega-3 fatty acids), Soy extracts (isoflavones), Green-tea preparations, Pomegranate extracts, Grape extracts
* Active malignancy
* Hepatitis virus or Human Immunodeficiency virus infections
* History of drug or alcohol dependency
* Cigarette smoking
* Psychiatric or neurological condition, preventing aware consent to the study and/or adherence to the study protocol

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary albumin-creatinine ratio | 3 month

SECONDARY OUTCOMES:
Change from baseline in urinary TNF-α | 3 month
Change from baseline in urinary TGF-β | 3 month
Change from baseline in fasting plasma glucose | 3 month
Change from baseline in blood lipid profile | 3 month
Change from baseline in hemoglobin A1C | 3 month
Change from baseline in urinary MDA | 3 month
Change from baseline in serum TNF-α | 3 month
Change from baseline in serum TGF-β | 3 month
Change from baseline in serum MDA | 3 month
Change from baseline in estimated GFR | 3 month
Change from baseline in serum creatinine | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Ghazal Vessal, PharmD, PhD, Study Director — Shiraz University of Medical Sciences, Faculty of Pharmacy; Mohammad Mehdi Sagheb, MD, Study Chair — Shiraz University of Medical Sciences; Jamshid Roozbeh, MD, Principal Investigator — Shiraz University of Medical Sciences, Nephrology Urology Research Center; Mohammad Kazem Fallahzadeh Abarghouei, M.D., Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Motahari Clinic, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Fallahzadeh MK, Dormanesh B, Sagheb MM, Roozbeh J, Vessal G, Pakfetrat M, Daneshbod Y, Kamali-Sarvestani E, Lankarani KB. Effect of addition of silymarin to renin-angiotensin system inhibitors on proteinuria in type 2 diabetic patients with overt nephropathy: a randomized, double-blind, placebo-controlled trial. Am J Kidney Dis. 2012 Dec;60(6):896-903. doi: 10.1053/j.ajkd.2012.06.005. Epub 2012 Jul 7. PMID 22770926